CLINICAL TRIAL: NCT01625234
Title: Phase 1/2, First-in-Human, Dose-Escalation Study of X-396 (Ensartinib) in Patients With Advanced Solid Tumors and Expansion Phase in Patients With ALK-positive Non-Small Cell Lung Cancer
Brief Title: Phase 1/2 Study of X-396, an Oral ALK Inhibitor, in Patients With ALK-positive Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Xcovery Holdings, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: X396-CLI-101
Record Dates: First submitted 2012-06-15; First posted 2012-06-21 (Estimated); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: Advanced Solid Tumors; Non-small Cell Lung Cancer
Keywords: Cancer; Tumors; ALK; NSCLC; Advanced Malignancies; Carcinoma, Non-Small-Cell Lung; Inflammatory Myofibroblastic Tumors
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms | interventions — ensartinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phase I: X-396 (ensartinib) (Experimental): Dose escalation starting at 25 mg, oral once or twice a day, 28-day cycle. Number of Cycles: until progression or unacceptable toxicity develops
  Interventions: Drug: Phase I: X-396 (ensartinib)
- Phase II: X-396 (ensartinib) (Experimental): RP2D 225mg stratified based on prior treatment and CNS activity
  Interventions: Drug: Phase II: X-396 (ensartinib)

INTERVENTIONS:
Drug: Phase I: X-396 (ensartinib) — Oral, ALK inhibitor
  Other Names: ensartinib
  Arms: Phase I: X-396 (ensartinib)
Drug: Phase II: X-396 (ensartinib) — Expanded Cohort
  Other Names: ensartinib
  Arms: Phase II: X-396 (ensartinib)

SUMMARY:
This is the first human study to use X-396 (ensartinib), a drug being developed for treatment of advanced cancers. The initial purpose of the study is to determine the largest amount of X-396 that can be safely given to humans (the maximum tolerated dose). Once the recommended Phase 2 dose has been determined, an expansion phase will assess the preliminary anti-tumor activity of X-396 in ALK-positive non-small cell lung cancer. The study will also provide early information on how the body handles the drug (pharmacokinetics) and on the efficacy of X-396.

DETAILED DESCRIPTION:
This is the first study of X-396 (ensartinib) in humans and the investigational drug will be given as a once or twice daily oral dose in 28 day cycles until there is disease progression or unacceptable safety issues. X-396 will be given to small groups of patients (1 - 6) at each dose level and the patients will be observed to see if there are any adverse safety effects. As long as there are no unacceptable safety issues after 28 days, the dose of X-396 will be increased for the next group of patients. This process will continue until the maximum tolerated dose (MTD) of X-396 is reached. Once the MTD is reached, up to 170 additional patients will also be given X-396 to further determine the activity of X-396 in patients with ALK-positive non-small cell lung cancer. These additional patients will be enrolled in the following expansion cohorts: ALK TKI-naïve patients, patients that progressed on crizotinib, patients that progressed on one or more 2nd generation ALK TKIs (patients may or may not have also received prior crizotinib), including patients with asymptomatic CNS metastases.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed diagnosis of advanced solid tumor malignancy. Patients may be ALK TKI-naive or may have received prior crizotinib and/or second generation ALK TKIs. In addition, patients with a known ALK 1198 mutation will be allowed.

   -For the expanded cohort portion of the study, patients must have NSCLC with ALK genomic alterations; however, patients will be allowed to enroll based on local FDA-approved ALK results.
2. Eastern Cooperative Group ECOG) Performance Status score of 0 or 1.
3. Ability to swallow and retain oral medication.
4. Adequate organ system function.
5. Patients with treated or untreated asymptomatic CNS metastases may be allowed to enroll.
6. Male patients willing to use adequate contraceptive measures.
7. Female patients who are not of child-bearing potential, and female patients of child-bearing potential who agree to use adequate contraceptive measures.
8. Patients must be ≥ 18 years of age.
9. Patients must have measurable or evaluable disease for the dose escalation portion of the study and measurable disease for the expanded cohort portion of the study (except for patients in the CNS metastases and leptomeningeal cohorts).
10. Willingness and ability to comply with the trial and follow-up procedures.
11. Ability to understand the nature of this trial and give written informed consent.

Exclusion Criteria:

1. Patients currently receiving cancer therapy.
2. Use of an investigational drug within 21 days or 5 half-lives (whichever is shorter) prior to the first dose of X-396. A minimum of 10 days between treatment and X-396 and 2 days between ALK TKI and X-396.
3. Any major surgery, radiotherapy, or immunotherapy within the last 21 days (focal radiation does not require a washout period; ≥4 weeks for WBRT). Chemotherapy regimens with delayed toxicity within the last 4 weeks. Chemotherapy regimens given continuously or on a weekly basis with limited potential for delayed toxicity within the last 2 weeks.
4. Prior stem cell transplant.
5. Patients with a known allergy or delayed hypersensitivity reaction to drugs chemically related to X-396 (e.g., crizotinib) or to the active ingredient of X-396.
6. Patients with primary CNS tumors are ineligible.
7. Patients receiving CYP3A substrates with narrow therapeutic indices, strong CYP3A inhibitors, and strong CYP3A inducers.
8. Concomitant use of herbal medications at least 7 days prior to the first dose of study drug and throughout participation in the trial.
9. Females who are pregnant or breastfeeding.
10. Presence of active gastrointestinal (GI) disease or other condition that will interfere significantly with the absorption, distribution, metabolism, or excretion of X-396.
11. Clinically significant cardiovascular disease.
12. Patients who are immunosuppressed (including known HIV infection), have a serious active infection at the time of treatment, have known hepatitis C, or have any serious underlying medical condition that would impair the ability of the patient to receive protocol treatment.
13. Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol.
14. Concurrent condition that in the investigator's opinion would jeopardize compliance with the protocol or would impart excessive risk associated with study participation that would make it inappropriate for the patient to be enrolled.
15. Inability or unwillingness to comply with study and/or follow-up procedures outlined in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2012-06; Primary Completion 2020-09-17 (Actual); Study Completion 2020-09-17 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | 12 months
  To evaluate the safety/tolerability of X-396 (ensartinib) and determine the maximum tolerated dose (MTD) of X-396 as a single agent.

SECONDARY OUTCOMES:
Plasma Concentrations (Cmax, Tmax, AUC, half-life) | 18 months
  To characterize the preliminary pharmacokinetics including Cmax, Tmax, AUC, half-life of X-396 given as a single agent
Preliminary Tumor Response | 18 months
  To explore the preliminary clinical tumor response after treatment with X-396 (ensartinib) given as a single agent.

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - City of Hope National Med Ctr, Duarte, California
  - UCSD Moores Cancer Center, La Jolla, California
  - University of Southern California Norris Comprehensive Cancer Center, Los Angeles, California
  - Stanford University, Stanford, California
  - Moffitt Cancer Center, Tampa, Florida
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - New York University Langone Medical Center, New York, New York
  - Providence Portland Medical Center, Portland, Oregon
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Vanderbilt University, Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Wisconsin Carbone Cancer Ctr, Madison, Wisconsin

REFERENCES:
- [Background] Lovly CM, Heuckmann JM, de Stanchina E, Chen H, Thomas RK, Liang C, Pao W. Insights into ALK-driven cancers revealed through development of novel ALK tyrosine kinase inhibitors. Cancer Res. 2011 Jul 15;71(14):4920-31. doi: 10.1158/0008-5472.CAN-10-3879. Epub 2011 May 25. PMID 21613408
- [Result] Horn L, Infante JR, Reckamp KL, Blumenschein GR, Leal TA, Waqar SN, Gitlitz BJ, Sanborn RE, Whisenant JG, Du L, Neal JW, Gockerman JP, Dukart G, Harrow K, Liang C, Gibbons JJ, Holzhausen A, Lovly CM, Wakelee HA. Ensartinib (X-396) in ALK-Positive Non-Small Cell Lung Cancer: Results from a First-in-Human Phase I/II, Multicenter Study. Clin Cancer Res. 2018 Jun 15;24(12):2771-2779. doi: 10.1158/1078-0432.CCR-17-2398. Epub 2018 Mar 21. PMID 29563138